CLINICAL TRIAL: NCT03645408
Title: The Effects of Exenatide, a GLP-1 Agonist, on Alcohol Self-Administration in Heavy Drinkers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to COVID-19 hospital-wide policies halting recruitment
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-38015; R21AA027332-01 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Alcohol Use Disorder
Keywords: exenatide; alcohol craving; alcohol consumption
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Exenatide; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled, crossover design trial that tested the effect of exenatide on alcohol self-administration and craving following a priming dose of alcohol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Nursing staff at the general Clinical Research unit were not blinded to the study medication. These nurses' only role in the study was providing injections of the study drug. All other staff were blinded to medication assignments. The sham injection was a needlestick using the exenatide multi-dose syringe with no drug injected. Note that the volume of fluid injected for a 5mcg dose was only .08ml. It is not expected that subjects would sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind. The individual who administered medication did not participate in subject evaluation to maintain the study blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide then Placebo (Experimental): This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this arm received a 5 mcg dose of immediate release exenatide on the day of the first alcohol self-administration trial. The 5mcg dose of exenatide was approved as the first dose administered to patients at the start of their treatment with this drug for FDA-approved indications. Subjects in this arm then received a sham injection on the day of the second alcohol self-administration trial. The sham injection was a needle stick using a syringe with no drug injected. Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
  Interventions: Drug: Exenatide; Other: Sham injection
- Placebo then Exenatide (Experimental): This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this arm received a sham injection on the day of the first alcohol self-administration trial. The sham injection was a needle stick using a syringe with no drug injected. Subjects in this arm then received a 5 mcg dose of immediate release exenatide on the day of the second alcohol self-administration trial. The 5mcg dose of exenatide was approved as the first dose administered to patients at the start of their treatment with this drug for FDA-approved indications. Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
  Interventions: Drug: Exenatide; Other: Sham injection

INTERVENTIONS:
Drug: Exenatide — Subject received an injection of 5 mcg of immediate release exenatide.
  Other Names: Byetta
Other: Sham injection — Subjects received a sham injection with no study drug.
  Other Names: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, crossover design trial was used to test the effect of exenatide on alcohol self-administration and craving following a priming dose of alcohol. The specific objective of this research was to determine whether exenatide has effects on alcohol consumption.

DETAILED DESCRIPTION:
This proposal was intended to answer the call for accelerating drug development by exploring the potential of a glucagon-like peptide-1 (GLP-1) agonist, exenatide, as a candidate medication for the treatment of Alcohol Use Disorder. There is now substantial preclinical evidence that GLP-1 agonists can attenuate behaviors that model both the consumption and seeking of several commonly abused substances including alcohol, cocaine, and nicotine. This study was intended to accelerate medication development for Alcohol Use Disorder by testing a commercially-available and well-tolerated agent at a fraction of the cost of new drug discovery. None of the FDA-approved Alcohol Use Disorder medications or off-label Alcohol Use Disorder medications target this GLP-1 pathway, making exenatide a promising compound for Alcohol Use Disorder drug development.

The primary aim of this study was to test the effects of exenatide on alcohol self-administration and craving among heavy drinkers. In this within-subjects crossover design, 3 heavy drinkers were randomized to exposure order (exenatide or sham injection) prior to completing two alcohol self-administration trials. Subjects received a priming drink of alcohol and had access to 8 drinks over a 2-hour period. The investigators anticipated that subjects would consume less alcohol following the administration of exenatide compared to when they received a sham injection. Significant exenatide-induced reductions in drinking would be considered to be an indication that this drug may have value as an Alcohol Use Disorder medication. This study may provide a rationale for phase II randomized controlled trials testing exenatide with a treatment-seeking Alcohol Use Disorder population. These results may also help to spur further clinical investigation of the effects of exenatide and other available GLP-1 agonists on the factors implicated in the regulation of alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

1. 21-55 years of age.
2. Able to verify age with a state or federal picture identification.
3. Exceeds safe weekly drinking limits [4 standard drink units (SDUs) for women or 21 SDUs for men per week]
4. Reports at least one episode of binge drinking (>3 SDUs for women, >4 SDUs for men) an average of once per week in the four weeks prior to baseline screening.
5. Meets Diagnostic And Statistical Manual Of Mental Disorders, Fifth Edition (DSM-5)criteria for mild alcohol use disorder or greater severity.

Exclusion Criteria:

1. Seeking treatment for alcohol problems.
2. Clinical Institute Withdrawal Assessment at ≥10
3. DSM-5 diagnosis of current major depression, bipolar disorder, schizophrenia, bulimia/anorexia, dementia, or a substance use disorder other than alcohol, nicotine, marijuana or caffeine.
4. If female, pregnant, nursing, have plans to become pregnant.
5. If female, does not agree to use an accepted form of birth control.
6. Has a medical contraindication to the use of exenatide.
7. Has medical or mental condition for which further alcohol exposure at the planned dose range would be contraindicated.
8. Current risk of suicidality (MINI suicidality score greater than 8 (low risk) or Yes to the ideation question #4 of the C-SSRS).
9. BMI is less than 18 or greater than or equal to 30.
10. History of diabetes.
11. Baseline hemoglobin A1c ≥ 6.5%
12. Baseline non fasting glucose >200
13. Significantly elevated serum lipase levels.
14. Impaired renal function (GFR <80 mL/min).
15. Pancreatitis, gastroparesis or other severe gastrointestinal disease.
16. Has had gastric bypass surgery
17. Subject is currently taking warfarin.
18. Has received alcohol counseling or other non-pharmacologic intervention to treat AUD in the past 90 days.
19. Has taken medications that are used to treat alcohol use disorder (AUD) in the past 90 days.
20. Subjects with a history of thyroid cancer or other thyroid disease.
21. Has urine toxicology results positive for cocaine, opioids, amphetamines, buprenorphine, methadone, or methamphetamines.
22. Prior history of anaphylaxis or angioedema with another GLP-1 receptor agonist.
23. Prior use of exenatide
24. Liver function values AST or ALT are twice the normal limit
25. Unable to comfortably abstain from nicotine for a period of 8 hours.
26. Has Chronic obstructive pulmonary disease (COPD), history of solid organ transplant, sickle cell disease, severe heart disease or other health condition for which exposure to COVID-19 represents an unreasonable risk as determined by the study staff physician using accepted COVID-19 guidance (e.g. Centers for Disease Control, etc.).
27. Subject has prior history of Drug-induced thrombocytopenia

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Devine, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Psychiatry Research Center, Clinical Studies Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 subjects were consented, 3 subjects were randomized, and 3 subjects completed the study.
Groups:
- Exenatide Then Placebo: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this arm received a 5 mcg dose of immediate release exenatide on the day of the first alcohol self-administration trial. The 5mcg dose of exenatide was approved as the first dose administered to patients at the start of their treatment with this drug for FDA-approved indications. Subjects in this arm then received a sham injection on the day of the second alcohol self-administration trial. The sham injection was a needle stick using a syringe with no drug injected. Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
  Sham injection: Subjects will have a sham injection with no study drug
Period: Overall Study
Arm/Group | Exenatide Then Placebo | Placebo Then Exenatide
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Then Placebo | Placebo Then Exenatide | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (0) | 23.5 (2.12) | 30.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Greater Boston, MA Area
  participants
    United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption
Description: Alcohol consumption was measured by using a graduated cylinder to determine the amount of alcohol given to the subject that was not consumed. The amount not consumed was then subtracted from the total amount of alcohol served to the subject in order to calculate the amount consumed. This outcome was measured in standard drink units (SDUs). A standard drink contains approximately 0.6 fluid ounces of pure alcohol.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: standard drink units (SDUs)
Groups:
- Exenatide Injection: Subjects received a 5 mcg dose of immediate-release exenatide on the day of the alcohol self-administration trial.
  This is a within subjects design study in which each subject received both study drug and sham injection (placebo). Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
- Sham Injection (Placebo): Subjects received a sham injection on the day of the alcohol self-administration trial.
  This is a within subjects design study in which each subject received both study drug and sham injection (placebo). Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
Arm/Group | Exenatide Injection | Sham Injection (Placebo)
Number analyzed (Participants) | 3 | 3
standard drink units (SDUs) | 0.93 (0.87) | 2.78 (2.66)

ADVERSE EVENTS:
Time Frame: Up to 38 days
Description: The primary risks of this study were risks related to taking study medication, loss of confidentiality, discomfort with study procedures, overconsumption of alcohol, and interference with efforts for recovery from alcohol use disorder. The protocol was designed to minimize risk to subjects.
Groups:
- Exenatide: Subjects received a 5 mcg dose of immediate-release exenatide on the day of the alcohol self-administration trial.
  This is a within subjects design study in which each subject received both study drug and sham injection (placebo). Note that the volume of fluid injected for a 5mcg dose is so small that subjects would not sense this volume of fluid (or lack thereof) during the injection. Subjects were shielded from seeing the injection to maintain the blind.
Arm/Group | Exenatide | Sham Injection (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=3) | Sham Injection (Placebo) (N=3)
Pre-drug injection anxiety (General disorders) | 0 (0) | 1 (1) — Subject experienced anxiety prior to receiving the injection of the study drug.
Nausea (General disorders) | 1 (1) | 0 (0) — Subject experienced mild nausea after receiving the study drug. This a known side effect of the study drug.

LIMITATIONS AND CAVEATS:
The small sample size reflects the early termination of the research which was halted due to Covid 19 precautions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03645408/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT03645408/ICF_001.pdf